CLINICAL TRIAL: NCT07135713
Title: Electrocardiographic Changes Associated With Epilepsy in Children Attending Assiut University Children's Hospital
Brief Title: Electrocardiographic Changes Associated With Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samaan Rezk Gad El Kariem, Resident Doctor, Department of Pediatrics, Assiut University Children's Hospital, Assiut University
Other Study IDs: Electrocardiographic Changes
Record Dates: First submitted 2025-07-18; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: ECG Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Identify and characterize electrocardiographic (ECG) changes occurring during the post-ictal phase of epileptic seizures. Evaluate the duration and severity of post-ictal ECG abnormalities. Assess the correlation between ECG changes and seizure type, duration, and severity. Explore the association of ECG changes with patient demographics

DETAILED DESCRIPTION:
Epilepsy is a chronic disease triggered by increased impulsiveness of nerve cells in the brain and may require a lifelong treatment. Epilepsy is confirmed by two or more unprovoked seizures in more than 24 hours, Febrile Convulsion (FC) is another type of seizure occurring due to fever over 38 °C without a history of convulsion, CNS infection, electrolyte imbalance, metabolic disorder, intoxication, and trauma

. Epilepsy is one of the most common neurological conditions which occurs in approximately 0.5-1% of children worldwide. However, it is not a disease entity but a syndrome of symptoms that can occur against various morphological and metabolic changes in the brain. One of the symptoms of epilepsy is epileptic seizures, i.e., temporary bioelectrical disturbances in the nerve cells of the brain . The simplified classification of epileptic seizures distinguishes between generalized seizures and partial (focal) seizures, depending, among other things, on the area of the brain where the discharges occur. Determination of the epileptic syndrome, i.e., the specific set of seizure types and electroencephalographic and imaging features, is the final stage of diagnosis . The cause of epilepsy is very often not recognized, and for this reason the diagnosis should be based on a thorough history of the patient, witnesses to the seizures, electroencephalogram (EEG) studies, and structural and functional neuroimaging of the central nervous system . One of the most dangerous changes occurs due to epileptic seizures are cardiovascular changes, which may result in sudden unexpected death in epileptic patients. Moreover, seizure leads to disturbance in cardiac functions and resulting in syncopal events, notablygeneralized convulsive seizures, put the cardiovascular system on strain, which may promote cardiac complications such as cardiac arrhythmias, cardiomyopathy, and myocardial infarction . A significant proportion of patients saw a rise in cardiac necrosis and dysfunction indicators after protracted convulsions, which might signal the beginning of myocardial damage Relevant abnormalities like prolonged QTc interval or cardiac block can be detected by a 12-lead ECG, which is an inexpensive test. Hypocalcemia as a cause of convulsions can be identified on an electrocardiogram (ECG) by a QTc prolongation due to a ST segment elongation, the severity of which is inversely related to the serum calcium level . Electrocardiographic changes in patients with drug-resistant epilepsy discovered that patients with epilepsy had significantly longer mean PR intervals, shorter mean QRS durations, shorter mean QTc intervals, and longer corrected QT interval dispersion than subjects without epilepsy . Cardiac electrical and functional abnormalities also have been described in children with epilepsy suggesting that the epileptic heart may affect pediatric patients. Implicit in the concept of the epileptic heart is that the epilepsy chronicity may be associated with an increased risk of developing cardiovascular complications. To date, only a few studies with small numbers of patients or highly selective populations have demonstrated the associations between cardiac alterations and longstanding epilepsy . ECG changes are commonly observed in epilepsy which make ECG a promising candidate to monitor seizure risk. Most ECG research in this domain has focused on heart rate-related changes. However, several studies have identified a range of other peri-ictal ECG parameter changesthat may potentially prove useful for seizure detection and forecasting.

ELIGIBILITY:
Inclusion Criteria:

1. Children from 1 year to 18 year are diagnosed with epilepsy.
2. Routine EEG.

Exclusion Criteria:

1. Known pre-existing cardiac conditions e.g arrhythmias, heart failure.
2. Current use of medications significantly affecting ECG.
3. Other causes of convulsion:hypoglycemia,hypernatriemia.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Eighty (80) children with epilepsy will be included in this study during the period from October 2025 to October 2026. Sample size was calculated by Open Epi Info version 3
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Out come measure | Baseline (immediate post-ictal phase)
  Title: Prevalence of Post-Ictal Electrocardiographic (ECG) Abnormalities Description: The proportion of participants who experience post-ictal ECG abnormalities, including sinus tachycardia, bradycardia, QT/QTc interval changes, ST-T segment changes, atrial/ventricular ectopy, or conduction blocks. Assessment will be performed using a standard 12-lead electrocardiogram (ECG).
  Unit of Measure: Percentage of participants

REFERENCES:
- [Background] Katyayan A, Diaz-Medina G. Epilepsy: Epileptic Syndromes and Treatment. Neurol Clin. 2021 Aug;39(3):779-795. doi: 10.1016/j.ncl.2021.04.002. PMID 34215386
- [Background] Ibrahim A, Megahed A, Salem A, Zekry O. Impact of Cardiac Injury on the Clinical Outcome of Children with Convulsive Status Epilepticus. Children (Basel). 2022 Jan 18;9(2):122. doi: 10.3390/children9020122. PMID 35204843
- [Background] Bastos F, Cross JH. Epilepsy. Handb Clin Neurol. 2020;174:137-158. doi: 10.1016/B978-0-444-64148-9.00011-9. PMID 32977874